CLINICAL TRIAL: NCT00885664
Title: Immune Reconstitution as a Determinant of Adverse Effects to New Antiretroviral Therapy in Persons With Advanced HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Abbott (Industry); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Carl J. Fichtenbaum, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDC 30
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: HIV Infections
Keywords: HIV; immune reconstitution; treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine; lopinavir-ritonavir drug combination; Lopinavir; Ritonavir

STUDY DESIGN:
Intervention Model Description: All participants received truvada and kaletra in this trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Truvada/Kaletra CD4<100 (Other): All participants were treated but at baseline by design were divided based upon their CD4 count at baseline measurement. Group with CD4<100 cells/cu mm
  Interventions: Drug: Truvada (tenofovir/emtricitabine); Drug: Kaletra (lopinavir/ritonavir)
- Truvada/Kaletra CD4>/=100 (Other): All participants were treated but at baseline by design were divided based upon their CD4 count at baseline measurement. Group with CD4>/=100 cells/cu mm
  Interventions: Drug: Truvada (tenofovir/emtricitabine); Drug: Kaletra (lopinavir/ritonavir)

INTERVENTIONS:
Drug: Truvada (tenofovir/emtricitabine) — Tenofovir/emtricitabine fixed dose combination once daily
  Other Names: Truvada
Drug: Kaletra (lopinavir/ritonavir) — Lopinavir/ritonavir 400/100 mg twice daily
  Other Names: Kaletra

SUMMARY:
The purposes of this study are:

1. To understand whether the use of HIV therapy in persons with more advanced HIV disease results in greater side effects.
2. To determine whether these side effects can be related to greater activation of the immune system.

DETAILED DESCRIPTION:
1. To compare the incidence and severity of self-reported symptoms in persons with CD4 counts <100 cells/mm3 versus those with CD4 counts ≥ 100 cells/mm3 who are initiating antiretroviral therapy.
2. To determine the relationship between self-reported symptoms and levels of T cells, HIV RNA, activation marker cytokines including TNF-α, IFN-γ, IL-2, IL-4, IL-6, IL-10 and other cytokines as measured before and after the initiation of antiretroviral therapy.
3. To determine the relationship between antiretroviral drug trough levels (estimated drug concentrations) and the incidence and severity of self-reported symptoms in persons initiating antiretroviral therapy.
4. To determine the relationship between adverse events and immunological status as evidenced by lymphocyte counts and activation marker cytokine levels.
5. To determine the relationship between clinical events and immunological status as evidenced by lymphocyte counts and activation marker cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Diagnosis of HIV infection.
3. Naive to antiretroviral therapy OR no use of antiretrovirals for ≥ 6 months.

Exclusion Criteria:

1. Blinded drug treatment.
2. Active untreated serious infection within 14 days of enrollment that in the opinion of the investigator would affect the subject's participation and/or safety in the study.
3. Known resistance to proposed new HIV regimen or components of regimen.
4. Requirement for drug therapy with known contraindication with proposed new antiretroviral therapy (see Prohibited and Precautionary Medications below)
5. Pregnancy or breast feeding.
6. Liver enzyme abnormalities on screening. Patients who have symptomatic Grade 3 elevations of total bilirubin, AST, ALT, or alkaline phosphatase or Grade > 3 elevations of total bilirubin, AST, ALT, or alkaline phosphatase will be excluded. Patients who have asymptomatic grade 3 elevations of total bilirubin, AST, ALT, or alkaline phosphatase may be included in the study at the discretion of the primary physician in consultation with the principal or senior investigator. Patients with grade 3 elevations of liver function tests who are co-infected with hepatitis B or hepatitis C may be included in the study at the discretion of the primary care physician in consultation with the primary or senior investigator provided that they do not have signs or symptoms of clinical hepatitis. Signs of clinical hepatitis include: icterus, abdominal tenderness and hepatosplenomegaly. Symptoms of clinical hepatitis include: fever, abdominal pain, anorexia, nausea, vomiting, fatigue, malaise, and myalgia.
7. Decreased creatinine clearance at the time of screening. Patients with a creatinine clearance of <50mL/min as calculated by the Cockcroft-Gault method should be excluded from study entry. The Cockcroft-Gault method is defined on page 33.
8. Other Grade ≥3 lab abnormalities. For any other laboratory abnormalities of grade 3 or higher, patients may be included or excluded from the study at the discretion of the primary care physician in consultation with the primary or senior investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-10; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Fichtenbaum, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati AIDS Clinical Trials Unit, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Academic HIV practice from October 2005 through March 2009.
Groups:
- Truvada/Kaletra: All participants received the same treatment. This was a single arm study.
Period: Overall Study
Arm/Group | Truvada/Kaletra
Started | 60
Completed | 48
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- Truvada/Kaletra CD4<100: Group with CD4 lymphocyte count less than 100 cell/cu mm treated with truvada/kaletra
- Truvada/Kaletra CD4>/=100: Group with CD4 lymphocyte count greater than or equal to 100 cell/cu mm
- Total: Total of all reporting groups
Arm/Group | Truvada/Kaletra CD4<100 | Truvada/Kaletra CD4>/=100 | Total
Number analyzed (Participants) | 26 | 34 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 34 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [36 to 49] | 37 [33 to 43] | 39.5 [20 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 24 | 31 | 55

OUTCOME MEASURES:

1. Primary Outcome: Symptom Score
Description: AIDS Clinical Trials Group Symptom Summary Score (20 item scale with severity from 0-4); Severity scale, 0=absent, 1=is least severe and 4 is most severe. Minimum score = 0 units on scale. Maximum score = 80 units on scale.
Time Frame: Week 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- CD4<100: Subjects with baseline CD4 count < 100 cells/mm3
- CD4>/=100: CD4 count greater than or equal 100 cells/mm3
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
units on a scale | 10 [5 to 17] | 8 [6 to 13]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: SF-12 Physical Capacity Score
Description: Measure of physical function out of 100. Lower score means less physical capacity.
Time Frame: 4 weeks
Population: Those with lower CD4 at baseline compared to those with a higher CD4 count.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
units on a scale | 43 [35 to 52] | 54 [46 to 55]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: SF-12 Mental Capacity Score
Description: Measure of mental functioning where lower is better out of a scale of 100.
Time Frame: 4 weeks
Population: lower CD4 count at baseline compared to higher CD4 counts
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
score on a scale | 46 [31 to 57] | 50 [39 to 54]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: IL-1 Beta
Description: Cytokine IL-1 beta measurement by Luminex multiplex assay in picograms/mL, dynamic range 0.13-2000 pg/mL
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
pg/mL | 0.03 [0.03 to 0.45] | 0.03 [0.03 to 0.03]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: IL-4
Description: Interleukin-4 measured by Luminex multiplex assay in picograms/mL, dynamic range 0.13-2000 pg/mL
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
pg/mL | 0.07 [0.07 to 0.73] | 0.07 [0.07 to 1.47]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: IL-6
Description: Interleukin 6 measured by Luminex multiplex assay in picograms/mL, dynamic range 0.13-2000 pg/mL
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
pg/mL | 4.41 [2.11 to 8.46] | 4.01 [1.94 to 17.43]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: IL-7
Description: Interleukin 7 measured by Luminex multiplex assay in picograms/mL, dynamic range 0.13-2000 pg/mL
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
pg/mL | 17.50 [12.36 to 24.30] | 10.53 [6.98 to 16.84]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: IL-8
Description: Interleukin 8 measured by Luminex multiplex assay in picograms/mL, dynamic range 0.13-2000 pg/mL
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
pg/mL | 7.58 [5.83 to 9.83] | 5.18 [4.22 to 7.06]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: IL-10
Description: Interleukin 10 measured by Luminex multiplex assay in picograms/mL, dynamic range 0.13-2000 pg/mL
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
pg/mL | 21.32 [11.44 to 43.75] | 10.30 [6.93 to 24.25]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: TNF Alpha
Description: Tumor Necrosis Factor Alpha - measured by Luminex multiplex assay in picograms/mL, dynamic range 0.13-2000 pg/mL
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
pg/mL | 13.07 [8.55 to 20.58] | 9.07 [6.27 to 11.81]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: INF Gamma
Description: Interferon gamma measured by Luminex multiplex assay in picograms/mL, dynamic range 0.13-2000 pg/mL
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CD4<100 | CD4>/=100
Number analyzed (Participants) | 26 | 34
pg/mL | 2.24 [0.18 to 34.03] | 1.06 [0.15 to 4.74]
Statistical Analysis 1: Comparison: CD4<100 vs CD4>/=100; Test type: Superiority; p = 0.33, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All participants received the same treatment intervention, an FDA approved combination at the time of the study. Adverse events from the treatment are reported by CD4 group as determined at baseline <100 or greater than/equal to 100 cells/cu mm
Arm/Group | Truvada/Kaletra CD4<100 | Truvada/Kaletra CD4>/=100
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/34
Other Adverse Events (participants affected / at risk) | 26/26 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Truvada/Kaletra CD4<100 (N=26) | Truvada/Kaletra CD4>/=100 (N=34)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | NA — Onset of numbness, tingling and pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Truvada/Kaletra CD4<100 (N=26) | Truvada/Kaletra CD4>/=100 (N=34)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Fatigue (General disorders) | 24 (35) | 30 (47)
Fevers (General disorders) | 9 (9) | 5 (6)
Nausea (Gastrointestinal disorders) | 6 (9) | 4 (7)
Anxiety (Psychiatric disorders) | 3 (4) | 5 (7)
Night Sweats (General disorders) | 12 (16) | 10 (13)

LIMITATIONS AND CAVEATS:
Small study of 60 subjects. Some subjects did not complete all study visits limiting data available for each time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less